CLINICAL TRIAL: NCT06633614
Title: PREhabilitation of Frail Elderly PAtients Undergoing majoR surgEry at HOME (PREPARE-HOME) Using Smart Wearables: A Prospective Randomized Controlled Trial
Brief Title: PREhabilitation of Frail Elderly PAtients Undergoing majoR surgEry at HOME (PREPARE-HOME) Using Smart Wearables
Acronym: PREPARE@HOME
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Singapore General Hospital (Other)
Responsible Party: Principal Investigator, Ke Yuhe, Associate Consultant, Singapore General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 202410-01
Record Dates: First submitted 2024-09-30; First posted 2024-10-09 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2024-09

CONDITIONS: Frailty Syndrome
Keywords: Prehabilitation; Home-based; Perioperative Science; Wearable Technology
MeSH Terms: conditions — Frailty

STUDY DESIGN:
Intervention Model Description: This randomized controlled trial (RCT) will compare a prehabilitation program using wearable technology (swSEP) with standard preoperative care (uSEP) in elderly patients undergoing major abdominal surgery. Participants will be randomly assigned to either the intervention or control group, with stratification based on baseline physical function, surgical risk, and physiotherapist involvement. The intervention group will follow a personalized exercise program, remotely supervised via telemedicine, and monitored through a Fitbit Aspire 3 device. The control group will receive standard care without wearable technology. The trial will assess improvements in physical function, postoperative outcomes, and recovery at 4 weeks, aiming to determine the superiority of the prehabilitation program over standard care.
Masking Description: Blinding The investigators will not be blinded, as they will be responsible for prescribing the intervention bundle to participants in the intervention arm. However, hospital staff, including nurses and surgeons, will be blinded to the allocation of study arms. It is acknowledged that maintaining full blinding for the treating team in the postoperative period may be challenging, as study details could potentially be disclosed by participants who are not blinded. Efforts will be made to minimise such disclosures to preserve blinding where possible.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (No Intervention): Participants in the control group (uSEP) will receive the standard PREPARE program provided by the hospital, which includes preoperative physiotherapy education and a home exercise booklet (Supplementary Material: Educational Materials). This unsupervised, home-based programme consists of full-body aerobic, resistance, and respiratory exercises that participants will perform independently at home. Additionally, participants with a Maximal Inspiratory Pressure (MIP) of less than 100 cmH₂O will be given an Inspiratory Muscle Trainer (IMT) to enhance respiratory function.
- Intervention (Experimental): Participants in the intervention group (swSEP) will receive standard preoperative physiotherapy education in addition to a Fitbit Aspire 3 wearable device, which will track vital signs such as heart rate, physical activity, and sleep patterns. They will follow a personalised exercise program that is remotely supervised by a physiotherapist via telemedicine twice a week. The exercise regimen will consist of 20-minute sessions, at least three times per week, and will include three core components: strength training, aerobic exercise, and flexibility exercises. Strength training will involve 2-3 sets of full-body exercises, including combinations of upper body, lower body, and abdominal movements. Aerobic exercises will be performed at a minimum intensity of 40% of the participant's maximal heart rate (HRmax) for up to 20 minutes. Flexibility training will include six stretches, each held for 20 seconds and repeated twice, targeting the chest, arms, legs, and trunk.
  Interventions: Device: Supervised prehabilitation programme

INTERVENTIONS:
Device: Supervised prehabilitation programme — Participants will receive standard preoperative physiotherapy education along with a Fitbit Aspire 3 wearable device to track vital signs such as heart rate, physical activity, and sleep patterns. They will follow a personalized exercise program, supervised remotely by a physiotherapist via telemedicine twice a week. The program will include 20-minute sessions at least three times per week, focusing on strength training, aerobic exercises (at 40% of maximal heart rate), and flexibility exercises. Progress will be monitored through vital signs and workout data, with the physiotherapists adjusting the regimen as needed. Participants with low inspiratory pressure (MIP <100 cmH₂O) will receive an Inspiratory Muscle Trainer (IMT). Additionally, some participants may be provided with a portable cycle pedometer featuring adjustable resistance. To ensure safety, both participants and caregivers will receive a safety briefing, and a 24-hour emergency hotline.
  Other Names: swSEP
  Arms: Intervention

SUMMARY:
The goal of this clinical trial is to evaluate whether a prehabilitation program using wearable technology can improve physical function and postoperative outcomes in elderly patients (65 years or older) undergoing major elective non-cardiac surgery. The main questions it aims to answer are:

Does the prehabilitation program improve physical function, as measured by the 6-minute walk test (6MWT), from baseline to pre-surgery? Does the prehabilitation program reduce postoperative complications and enhance recovery? Researchers will compare participants who receive the prehabilitation program with wearable technology (intervention group) to those receiving standard preoperative care (control group) to see if the intervention results in greater improvements in physical function and postoperative outcomes.

Participants will:

Follow a personalized exercise program monitored remotely via telemedicine. Wear a Fitbit Aspire 3 device to track vital signs such as heart rate and physical activity.

Undergo assessments of physical function and quality of life before surgery.

DETAILED DESCRIPTION:
This clinical trial aims to investigate the effectiveness of a prehabilitation program using wearable technology to improve physical function and postoperative outcomes in elderly patients undergoing major elective non-cardiac surgery. The intervention group will receive a comprehensive preoperative rehabilitation program (swSEP) that includes personalized exercise regimens monitored via telemedicine and a wearable device (Fitbit Aspire 3) to track key physiological metrics such as heart rate, physical activity, and sleep patterns. The exercise program will consist of three components: strength training, aerobic exercises, and flexibility exercises. These sessions will be conducted three times per week, with adjustments made by the physiotherapist based on the participant's progress and vital sign responses.

Participants will be monitored closely through telemedicine check-ins twice per week to ensure adherence to the exercise program, address any challenges, and make modifications to the regimen as needed. In addition, all participants will undergo baseline functional assessments, including the 6-minute walk test (6MWT), 30-second sit-to-stand test (30sSTS), handgrip strength (HGS), and maximal inspiratory pressure (MIP), as well as nutritional and quality of life assessments using the MUST score and EQ-5D-5L questionnaire. These assessments will be repeated 1-3 days before surgery to evaluate any improvements in physical function.

The control group (uSEP) will receive standard preoperative care, which includes physiotherapy education and a home-based exercise booklet, but will not be provided with a wearable device or telemedicine supervision. Both groups will be monitored for postoperative outcomes, including the incidence of complications classified by the Clavien-Dindo system, hospital length of stay, ICU admissions, and hospital readmissions. Health-related quality of life (HRQoL) will also be measured at multiple time points.

Exploratory analyses will include postoperative recovery and resumption of physical activity at 12 weeks post-surgery, as well as heart rate variability (HRV) data from the wearable devices to assess physiological responsiveness to the prehabilitation program and its potential predictive value for postoperative outcomes. A qualitative interview study will be conducted concurrently to explore the barriers and facilitators of home-based prehabilitation from the perspectives of both patients and healthcare providers.

ELIGIBILITY:
Inclusion Criteria:

* Frail elderly patients aged 65 years or older.
* Scheduled to undergo major elective, non-cardiac surgery.
* Anticipated surgery duration of over two hours or expected blood loss greater than 500 mL.
* Frailty status with Edmonton Frail Scale (EFS) score of 6 or higher.
* Capacity to provide informed consent independently.
* Available at least two weeks before surgery to participate in the prehabilitation program.
* Ability to follow exercise instructions independently.
* Ownership of a smartphone with Bluetooth and cellular connectivity.

Exclusion Criteria:

* Severe comorbidities that interfere with participation in the exercise program (e.g., unstable angina, severe aortic stenosis, or uncontrolled arrhythmias).
* Cognitive impairments that prevent understanding or adherence to the intervention.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 190 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2027-09-30 (Estimated); Study Completion 2028-01-31 (Estimated)

PRIMARY OUTCOMES:
Change in Physical Function (6-Minute Walk Test) from baseline to before surgery. | baseline to 1-3 days pre-surgery.
  The primary outcome of this study will be the change in physical function from baseline to 1 to 3 pre-surgery, measured by the 6-minute walk test (6MWT).

SECONDARY OUTCOMES:
Functional assessments | Baseline to 1-3 days before the surgery
  Functional outcomes will encompass the 30-second sit-to-stand test (30sSTS) and handgrip strength (HGS) will be measured from baseline to 1-3 days before the surgery
Postoperative complications | Preoperative to up to 4 weeks after surgery.
  Postoperative complications will be categorised according to the ACS NSQIP postoperative complications criteria.
Health Services outcomes | Preoperative to up to 8 weeks after surgery.
  Health services outcomes, including hospital length of stay, intensive care unit (ICU) admissions, hospital readmissions, and associated healthcare costs, will also be recorded to assess the intervention's impact on healthcare resource utilisation. Health-related quality of life (HRQoL) will be evaluated using the EQ-5D-5L questionnaires before and 8 weeks after surgery.

IPD SHARING:
Plan to Share IPD: No
The participant data will be identifiable in this study, and is not passed by the ethics board to share the data.

REFERENCES:
- [Derived] Leong YH, Tay VYJ, Yang X, Tan CJ, Au-Yong PS, Sim JLX, Ng RRG, Ong MEH, Tan BPY, Abdullah HR, Ke Y. Prehabilitation of frail elderly PAtients undergoing majoR surgEry at HOME (PREPARE-HOME): a superiority parallel-group randomised controlled trial protocol evaluating smart wearable enhanced prehabilitation versus usual care. BMJ Open. 2025 Oct 23;15(10):e094986. doi: 10.1136/bmjopen-2024-094986. PMID 41130682